CLINICAL TRIAL: NCT01697046
Title: A Pilot Study of the Safety, Acceptability, Behavior Impact, and HIV Seroincidence Among High Risk Men Who Have Sex With Men With Access to Isentress 400 mg BID + Truvada Once Daily for Peri-exposure Chemoprophylaxis for HIV Infection Chemoprophylaxis for HIV Infection
Brief Title: A Pilot Study on Raltegravir, Tenofovir and Emtricitabine for Peri-exposure Prophylaxis for HIV Infection
Acronym: PERIEP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Projeto Praça Onze (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Mauro Schechter, MD, PhD, Projeto Praça Onze
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IIS# 39550
Record Dates: First submitted 2012-09-24; First posted 2012-10-02 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-09

CONDITIONS: Infection; HIV
Keywords: peri-exposure; chemoprophylaxis
MeSH Terms: conditions — Infections | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Isentress+Truvada (Experimental): All participants will receive the intervention
  Interventions: Drug: Truvada and Isentress

INTERVENTIONS:
Drug: Truvada and Isentress — Subjects with reported high-risk behavior (and anticipated future high-risk behavior) but no exposure in the immediate past will be the focus of this study.
  Participants will be prescribed raltegravir 400 mg BID + Truvada once daily. All study participants will receive a 4-days starter pack. Study participants will be instructed to start study drugs if they expect or experience an exposure of any mucous membrane (oral, urethral, anal) to semen. Subjects who expect or experience these exposures will be instructed to take 1 pill of Raltegravir 400mg and one pill of truvada, followed by a second dose of Raltegravir 12 hours later. From the second day onward, participants will be instructed to take Raltegravir 400 mg BID + Truvada once daily. The first dose should be taken no more than 6 hours before or 6 hours after the expected or actual exposure and continued for 28 days.

SUMMARY:
This will be a pilot, open label study involving 65 participants. All participants will be followed until seroconversion or until the last enrolled participant completes one year of follow-up, whichever happens first. Participant study number will be given at the screening visit, prior to inclusion in the study.

The chosen intervention and study regimen are based on the dynamics of viral infection and the pharmacokinetics of the study drugs. In order to inhibit reverse transcription nucleoside and nucleotide analogues need to be phosphorylated intracellularly. On the other hand, available data indicate that it takes approximately 10 hours between exposure and HIV viral integration, offering a window of opportunity for Raltegravir to block integration and thus prevent infection, given that this drug does not need to be metabolized to exert its effect. The intervention will be maintained for 4 weeks following exposure, in accordance with Brazilian and CDC guidelines for PEP.

DETAILED DESCRIPTION:
Subjects with reported high-risk behavior (and anticipated future high-risk behavior) but no exposure in the immediate past will be the focus of this study.

Participants will be prescribed raltegravir 400 mg BID + Truvada once daily. All study participants will receive a 4-days starter pack. Study participants will be instructed to start study drugs if they expect or experience an exposure of any mucous membrane (oral, urethral, anal) to semen. Subjects who expect or experience these exposures will be instructed to take 1 pill of Raltegravir 400mg and one pill of truvada, followed by a second dose of Raltegravir 12 hours later. From the second day onward, participants will be instructed to take Raltegravir 400 mg BID + Truvada once daily. The first dose should be taken no more than 6 hours before or 6 hours after the expected or actual exposure and continued for 28 days.

Enrolled subjects will also be instructed to report to the study site within 4 days of beginning study drugs to respond to a CASI questionnaire and to have blood taken. They will be instructed to return at the end of the 4-week chemoprophylaxis course for reevaluation and to be given another 4-day supply of medication. Under no circumstances will any participant be given a greater than 4 week supply of medication; all will be evaluated for toxicity and adherence following each course of chemoprophylaxis.

The study participants will be monitored closely for safety after each course of chemoprophylaxis and at the end of the trial. In addition, subjects will be instructed to immediately contact the site if they experience certain symptoms consistent with severe toxicity. At each evaluation a careful clinical history, physical examination, and laboratory assessment, including HIV serology, will be completed. Adherence will be estimated based on self-report and the use of pill counts. During each visit, subjects will be reminded of the need to not increase high-risk sexual behavior. HIV serology and response to a CASI questionnaire will be conducted monthly.

ELIGIBILITY:
Inclusion Criteria:

Individuals will be included in the clinical trial if they meet ALL of the following criteria:

* Male sex (at birth);
* Willing and able to provide written informed consent;
* Age 18 years or older;
* HIV-1-uninfected;
* Absence of signs or symptoms compatible with an acute viral disease
* Evidence of high risk for acquiring HIV-1 infection including any one of the following: 1) No condom use during the last receptive and/or insertive anal intercourse with a male HIV-positive partner or a male partner of unknown HIV status during the last 6 months; (2) anal intercourse with more than 4 male sex partners during the last 6 months; (3) exchange of money, gifts, shelter, or drugs for anal sex with a male partner during the last 6 months; (4) sex with a male partner and STI diagnosis during the last 6 months or at screening, or (5) sexual partner of an HIV-infected man with whom condoms are not consistently used.
* Adequate renal function
* Adequate hepatic function

Exclusion Criteria:

* Glycosuria or proteinuria
* Acute hepatitis B infection
* History of pathological bone fractures not related to trauma
* Active alcohol or drug use considered sufficient to hinder compliance with any study procedures
* At enrollment, has any other condition that, based on the opinion of the investigator or designee, would preclude provision of informed consent; make participation in the study unsafe; complicate interpretation of study outcome data; or otherwise interfere with achieving the study objectives

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Safety | 16 months
  Number and severity of adverse events

SECONDARY OUTCOMES:
HIV seroincidence | 16 months
  Rate of incidence of new infections

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Schechter, MD, PhD, Principal Investigator — Projeto Praça Onze
Locations (1):
- Monica Barbosa de Souza, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). Update: provisional Public Health Service recommendations for chemoprophylaxis after occupational exposure to HIV. MMWR Morb Mortal Wkly Rep. 1996 Jun 7;45(22):468-80. PMID 8622618
- [Background] Cardo DM, Culver DH, Ciesielski CA, Srivastava PU, Marcus R, Abiteboul D, Heptonstall J, Ippolito G, Lot F, McKibben PS, Bell DM. A case-control study of HIV seroconversion in health care workers after percutaneous exposure. Centers for Disease Control and Prevention Needlestick Surveillance Group. N Engl J Med. 1997 Nov 20;337(21):1485-90. doi: 10.1056/NEJM199711203372101. PMID 9366579
- [Background] Schechter M, do Lago RF, Mendelsohn AB, Moreira RI, Moulton LH, Harrison LH; Praca Onze Study Team. Behavioral impact, acceptability, and HIV incidence among homosexual men with access to postexposure chemoprophylaxis for HIV. J Acquir Immune Defic Syndr. 2004 Apr 15;35(5):519-25. doi: 10.1097/00126334-200404150-00010. PMID 15021317
- [Background] Grant, RM; Lama, JR; Anderson, PL; McMahan, V; Liu, AY; Vargas, L; Goicochea, P; Casapía, M; Guanira-Carranza, JV; Ramirez-Cardich, ME; Montoya-Herrera,O; Fernandez, T; Veloso, VG; Buchbinder, SP; Chariyalertsak, S; Schechter, M; Gail -Bekker, L; Mayer, KM; Kallas, EG; Amico, KR; Mulligan, K; Bushman, LR; Hance, TJ; Ganoza, C; Defechereux, P; Brian, P; Wang, F; McConnell, JJ; Zheng, JH; Lee, J; Rooney, JF; Jaffe, HS; Martinez, AI; Burns, DN; Glidden, DV. Pre-Exposure Chemoprophylaxis for HIV Prevention in Men who Have Sex with Men. New Eng J Med 2010; 363:2587-99.